CLINICAL TRIAL: NCT00513487
Title: Assessment of the Effects of Multiple Nasal Antigen Challenges With Dust Mite Allergen on Local and Systemic Allergic Inflammation and Bronchoreactivity in Subjects With Allergic Rhinitis Sensitive to House Dust Mite - a Feasibility and Site Evaluation Study
Brief Title: Effects of Multiple Nasal Exposures to House Dust Mite Allergen on Nasal and Body Inflammation and Airway Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CPJMR0052107
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; dust mites; IgE; IL-13; nasal; inflammation
MeSH Terms: conditions — Rhinitis, Allergic; Inflammation | interventions — Fluticasone; Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dust mite extract, Fluticasone, Methacholine — Dust mite extract, Fluticasone, Methacholine

SUMMARY:
This study will evaluate whether multiple nasal antigen challenges with dust mite allergen produces increases in nasal symptoms and local allergic inflammatory cells in the nose and the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking subjects with a history of allergic rhinitis consistent with dust mite allergy showing
* A positive skin prick test to dust mite at or within the 12 months before study start
* Demonstrate symptomatic worsening after graded nasal allergen challenge

Exclusion Criteria:

* Subjects found to be very sensitive to house dust mites (if the skin prick test produces a wheal of mean with a diameter greater than 11 mm).
* Presence of any respiratory disease other than a history of mild stable asthma not requiring regular treatment.
* Any known contraindications for methacholine challenge testing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-07; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score recorded at baseline, and at pre-challenge,15 mins, 30 mins,and at 1,2,3,4,8 hours | throughout the study

SECONDARY OUTCOMES:
Peak nasal inspiratory flow at time points of total nasal symptom score. Mechanistic markers during challenge days. Exhaled nitric oxide,forced expiratory vol in 1 second & airway resistance at baseline, first & last day | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Sydney, Australia